CLINICAL TRIAL: NCT05996562
Title: Study for Evaluation of Safety and Efficacy of Pulmonary Artery Denervation to TreatCombined Post- and Pre- Capillary Pulmonary Hypertension Associated With Chronic Heart Failure: A Pilot Study
Brief Title: Study for Evaluation of Safety and Efficacy of PADN to Treat Combined Post- and Pre- Capillary Pulmonary Hypertension Associated With Chronic Heart Failure（PADN-CpcPH-PILOT）
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pulnovo Medical (Wuxi) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pulnovo-CO-2023-01
Record Dates: First submitted 2023-07-25; First posted 2023-08-18 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Hypertension; Heart Failure
Keywords: Pulmonary Artery Denervation; PADN; Pulmonary Hypertension; Heart Failure
MeSH Terms: conditions — Hypertension, Pulmonary; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulmonary Artery Denervation (PADN) (Experimental)
  Interventions: Procedure: Pulmonary Artery Denervation

INTERVENTIONS:
Procedure: Pulmonary Artery Denervation — Contrast pulmonary artery (PA) angiography will be performed to localize the pulmonary artery bifurcation level and calculate the PA diameter. Once the anatomy deemed acceptable, the radiofrequency ablation catheter will be introduced into ostium of the left PA and the distal bifurcation area of the main PA.
  The catheter will be manoeuvred within the PA to allow energy delivery in a circumferential manner to ensure that the electrodes are tightly in contact with the endovascular surface. About three ablations at 45-55°C for 120 seconds each will be performed in ostium of the left PA and the distal bifurcation area of the main PA.

SUMMARY:
The goal of this pilot study is to evaluate the safety and efficacy of pulmonary artery denervation (PADN) in Combined Post- and Pre- Capillary Pulmonary Hypertension Associated with Chronic Heart Failure.

Participants who have received guideline-directed medical therapy (GDMT) according to 2022 AHA/ACC Guidelines for Heart Failure (HF) and have been clinically stable for at least 1 month, will be treated with PADN and followed for 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18, ≤85 years;
2. PH must be confirmed by RHC, defined as:

   1. Mean pulmonary arterial pressure (mPAP) >20mmHg, and;
   2. Pulmonary capillary wedge pressure (PCWP) >15mmHg, and；
   3. Pulmonary vascular resistance (PVR) > 2WU.
3. Chronic heart failure has been diagnosed at least 3 months before screening and have been treated on the GDMT according to 2022 AHA/ACC Guidelines for Heart Failure for at least 1 month;
4. Clinically stable HF for at least 1 month, defined as:

   1. No need of intravenous diuretics, inotropes or vasodilators, and
   2. Systolic blood pressure (SBP) ≥ 100 and < 160 mmHg, and
   3. Resting heart rate (HR) ≥ 50 bpm and <100 bpm (>110 bpm in presence of atrial fibrillation) on the day of the procedure.
5. NYHA class II-IVa;
6. 6MWD ≥ 100 m and ≤ 450 m;
7. NT-proBNP >125pg/mL (or BNP > 35pg/mL);
8. Understand and be willing to sign informed consent and be strictly willing to follow the protocol.

Exclusion Criteria:

1. Any of the following:

   1. Hypertrophic cardiomyopathy with left ventricular (LV) outflow tract obstruction and/or mitral valvular systolic anterior motion (SAM); or
   2. Pericardial disease; or
   3. Infiltrative or inflammatory myocardial disease; or
   4. Valvular heart disease with stenosis or with severe regurgitation; or
   5. Active endocarditis; or
   6. Symptomatic carotid stenosis, or TIA or stroke within 30 days prior to randomization; or
   7. Congenital heart disease; or
   8. Having received any revascularization, including coronary artery bypass grafting (CABG) or percutaneous coronary intervention (PCI) within 6 months prior to randomization; or anticipated to undergo coronary revascularization (CABG or PCI) within 6 months; or
   9. Artificial pacemakers, including single-chamber, dual-chamber and three-chamber pacemakers, have been implanted less than 6 months or are anticipated to be implanted within 6 months; or
   10. Anticipated to undergo ablation of atrial fibrillation within 6 months; or
   11. Anticipated to undergo heart valve surgery (valve replacement, valvuloplasty) within 6 months; or
   12. Listing for heart/heart-lung transplantation or anticipated to implant a ventricular assist device (VAD)
2. Received pulmonary arterial hypertension (PAH) targeted drugs within 1 month prior to randomization;
3. Anticipated to undergo any surgery within the next 6 months;
4. Cardiac index (CI) measured by RHC < 1.5L/min/m2;
5. Severe renal insufficiency (eGFR < 30mL/min/1.73m2 by MDRD formula);
6. Severe liver insufficiency (Child-Pugh classification B-C);
7. Platelet count < 50 × 109/L;
8. Life expectancy < 1 year;
9. Systemic inflammation or other disease requiring long-term use of glucocorticoids or immunosuppressants;
10. Active infection requiring oral or intravenous antibiotics;
11. Cannot tolerate warfarin, aspirin, clopidogrel, and any of GDMT medicines;
12. Body mass index (BMI) > 40 kg/m²;
13. Pregnant or lactating women, or planning to be pregnant within one year;
14. Participation in other clinical trials within 3 months prior to signing the informed consent;
15. Any other circumstances that investigators deemed inappropriate to participate in this trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-06-28 (Actual); Primary Completion 2026-01-15 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
6-minute walk distance (6MWD) difference | 6 months
  The primary endpoint is change in 6-min-walk distance (6-MWD) from baseline to 6months.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Santa Marta, Lisbon, Portugal